CLINICAL TRIAL: NCT00998712
Title: Gestational Diabetes Mellitus and Cardiovascular Disease: The Role of Vascular Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rhonda Bentley-Lewis, MD, Rhonda Bentley-Lewis, MD, MBA, MMSc, Brigham and Women's Hospital
Other Study IDs: 2009P001255
Record Dates: First submitted 2009-10-16; First posted 2009-10-20 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Gestational Diabetes Mellitus; Pregnancy
Keywords: gestational diabetes mellitus; pregnancy; cardiovascular disease risk
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Black women in the third trimester of a pregnancy complicated by gestational diabetes.
- 2: Black women in the third trimester of a normal, uncomplicated pregnancy.
- 3: White women in the third trimester of a pregnancy complicated by gestational diabetes.
- 4: White women in the third trimester of a normal, uncomplicated pregnancy.

SUMMARY:
The purpose of this research study is to look at whether there are differences in blood vessel function, risk for developing diabetes (high blood sugar), lipid (blood fat) levels, and levels of other blood markers between black women and white women who have or do not have gestational diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women of self-identified African descent (black) and European (white) ancestry,
* 18-40 years of age,
* Body mass index < 35 kg/m2
* History of regular menstrual cycles,
* Are currently pregnant and in third trimester of pregnancy (after 24 weeks gestational age)
* Have no pregnancy-associated complications to-date
* Are in good health free of hypertension, as well as thyroid, cardiac, or renal disease.

Exclusion Criteria:

* History of smoking
* Are taking potentially vasoactive medications

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Black and white women currently in the thrid trimester of a pregnancy complicated or uncomplicated by gestational diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2009-08; Primary Completion 2013-10 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
endothelial function | same day

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Massachusetts General Hospital, Boston, Massachusetts, United States